CLINICAL TRIAL: NCT01039870
Title: The Effect of Paravertebral Block Using a Multi-orifice Catheter on Preventing Acute and Chronic Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Young-Tae Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YTKim_PVB_Postthor Pain
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Acute Postthoracotomy Pain; Chronic Postthoracotomy Pain; Hypotension After Bolus Dose
Keywords: postthoracotomy pain
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVB (Experimental): Paravertebral block initiated at the later part of thoracotomy is used for postoperative pain control
  Interventions: Procedure: paravertebral block
- TEA (Active Comparator): Thoracic epidural block initiated before the surgical incision is used for postoperative pain control.
  Interventions: Procedure: thoracic epidural analgesia

INTERVENTIONS:
Procedure: paravertebral block — postoperative pain is controlled with local analgesics delivered via PVB
  Arms: PVB
Procedure: thoracic epidural analgesia — postoperative pain is controlled with local analgesics and fentanyl delivered via thoracic epidural catheter
  Arms: TEA

SUMMARY:
This study aims to evaluate the effect of the paravertebral block using a multi-lumen catheter on the incidence and severity of acute and chronic postthoracotomy pain compared to the thoracic epidural block.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving surgery through a thoracotomy incision

Exclusion Criteria:

* patients with cardiovascular disease
* patients with neurologic disease
* patients with contraindications to paravertebral block or epidural block
* patients with history of previous thoracotomy incision
* patients with pain at the expected incision site

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of acute postthoracotomy pain when moving | 24 hours after thoracotomy

SECONDARY OUTCOMES:
Incidence of chronic postthoracotomy pain | 6 months after thoracotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea